CLINICAL TRIAL: NCT06164288
Title: A Phase I Study to Evaluate the Safety and Efficacy of Human Amniotic Epithelial Stem Cell（hAESCs）Injection Treatment for the Patients With Refractory aGVHD After Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Safety and Efficacy Study of hAESCs Therapy for aGVHD
Acronym: aGVHD，hAESCs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAESCS-GVHD-101
Record Dates: First submitted 2023-11-21; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: GVHD,Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hAESCs injection (Experimental): Intravenous reinfusion of human amniotic epithelial cell injection, the number of injections is single
  Interventions: Drug: Human Amniotic Epithelial Stem Cell Injection

INTERVENTIONS:
Drug: Human Amniotic Epithelial Stem Cell Injection — The dose escalation is carried out according to the "3+3" ascending principle, and a total of 3 dose levels are set:
  1. Dose Level 1: 1×106 cells/kg;
  2. Dose Level 2: 2×106 cells/kg;
  3. Dose Level 3: 3×106 cells/kg; Note: In this study, if the maximum tolerated dose (MTD) is not explored at dose level 3 (3×106 cells/kg), it will be discussed by the Safety Review Committee (SRC) to decide whether to proceed with further dose escalation or expansion to 6 patients.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT), a process in which hematopoietic stem cells from a donor are injected into the recipient's body, are the treatment of choice for many hematologic malignancies. Graft-versus-host disease (GVHD) is a common and important complication after allogeneic HSCT. GVHD is a major obstacle to the success of HSCT treatment and a leading cause of death after HSCT treatment.

Hormone therapy is currently the standard treatment for aGVHD, i.e., the first-line treatment. However, 40%~50% of aGVHD cannot be controlled by hormone therapy, and additional therapeutic intervention is required. According to the National Comprehensive Cancer Network (NCCN) clinical practice guidelines for hematopoietic stem cell transplantation - pre-transplant recipient evaluation and management of GVHD (2021.V3), the recommended drugs for second-line treatment of grade II~IV aGVHD include: alemtuzumab, α-1 antitrypsin, antithymocyte globulin, basiliximab, calcineurin inhibitors, etanercept, extracorporeal photopheresis replacement therapy, infliximab, mammalian rapamycin target protein inhibitors, mycophenolate mofetil, Pentostatin, ruxolitinib, tocilizumab. Second-line treatment is based on retrospective data and there is no standard salvage therapy, which is reflected in the inconsistent treatment strategy for aGVHD across transplant centers.

One of the biological functions of hAESCs in amniotic membranes in vivo is to exert reproductive immunomodulatory effects and protect the fetus from rejection by the maternal immune system, so hAESCs have natural immunomodulatory functions. hAESCs have significant inhibitory effects on T cells, antigen-presenting cells (APCs), natural killer (NK) cells, macrophages, neutrophils, B cells and other immune cells associated with organ damage during the pathogenesis of aGVHD, and hAESCs have great potential in the treatment of aGVHD. Therefore, the sponsor developed hAESCs injections intended for the treatment of aGVHD.

The experimental drug in this study is hAESCs injection, which is intended to be used for the treatment of adult patients with grade III.~IV. refractory aGVHD after hematopoietic stem cell transplantation, and to explore the safety and preliminary efficacy of its treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or his/her guardian agrees to participate in this clinical trial and signs the informed consent form (ICF), indicating that he understands the purpose and procedures of this clinical trial and is willing to participate in the study;
2. Age≥ 18 years old, gender is not limited;
3. The first occurrence of refractory aGVHD diagnosed by modified Glucksberg criteria with an overall clinical score of III.~IV., if other causes can be ruled out by clinical diagnosis, etc., no biopsy is required to confirm the diagnosis, but the following conditions must be met at the same time:

   1. Patients with hematologic malignancies who have undergone transplantation from any hematopoietic stem cell source (bone marrow, peripheral blood, umbilical cord blood) and have myeloablative pretreatment before hematopoietic stem cell transplantation (acute lymphoblastic leukemia, chronic myeloid leukemia are preferred);
   2. Refractory aGVHD refractory to second-line drug therapy: those who have been treated with at least one second-line drug (anti-CD25 monoclonal antibody, ruxolitinib, etc.) after hormone resistance, and the aGVHD symptoms still progress or do not improve; Note: Hormone-resistant aGVHD is defined as disease progression (PD) (aGVHD exacerbation (at least one-grade increase in aGVHD in at least one target organ) (with or without improvement in aGVHD in other organs) within 3~5 days of intravenous methylprednisolone at an initial dose of 2 mg/kg/d or equivalent hormone therapy (with or without improvement in aGVHD in other organs) or no response (NR) within 5~7 days of treatment (no improvement or worsening in aGVHD severity in any target organ);14 days do not reach CR (disappearance of symptoms in all organs, i.e., aGVHD has an overall score of 0);
4. Eastern Cooperative Oncology Group (ECOG) score ≤ 2;
5. The functions of important organs meet the following conditions:

   1. Cardiac function: left ventricular ejection fraction ≥50%;
   2. Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3× upper limit of normal (ULN). If elevated AST and ALT are associated with aGVHD, AST and ALT ≤5× ULN;
   3. Renal function: creatinine (Cr) ≤1.5×ULN, or creatinine clearance (Ccr) ≥30 mL/min/1.73m2 (according to Cockcroft and Gault formula);
   4. Oxygen saturation at the end of the finger ≥92%;
6. When the subject or his/her spouse is a woman of childbearing age, the subject agrees to use effective contraception during the trial (the subject uses non-drug contraception).

Exclusion Criteria:

1. Being treated in another therapeutic clinical trial within 4 weeks before study treatment infusion;
2. Subjects with a history of other parenchymal organ transplantation;
3. Subjects who have received mesenchymal stem cell (MSC) or hAESCs therapy or other stem cell therapy (except hematopoietic stem cells) within 6 months before study treatment infusion;
4. Previous receipt of live virus or attenuated vaccination within 4 weeks before study treatment infusion;
5. Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) test higher than the upper limit of normal (if HBsAg, hepatitis B e antigen (HBeAg) and HBcAb are positive, HBV DNA test is not required and can be directly excluded); positive hepatitis C virus (HCV) antibody; positive human immunodeficiency virus (HIV) antibody; positive syphilis antibody test; Note: The above virological tests can accept laboratory test results within 1 month before enrollment.
6. Known allergic reaction to any of the ingredients used in the treatments involved in this study, including hAESCs, dimethyl sulfoxide (DMSO), and BAT);
7. Known lung diseases such as pulmonary fibrosis, interstitial lung disease, acute exacerbation of chronic obstructive pulmonary disease, active lung infection, etc., which are not controlled;
8. Severe hepatic vein occlusive disease;
9. Pregnant or lactating females;
10. Subjects judged by the investigator to have difficulty completing all visits or operations required by the study protocol (including follow-up periods), or insufficient compliance with participation in this study;
11. In the opinion of the investigators, the patient has any underlying or current medical or psychiatric condition that would interfere with the treatment and evaluation of the subject, including but not limited to medically controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg), uncontrolled infection, pulmonary hypertension, clinically significant (e.g., active) cardiovascular and cerebrovascular diseases such as cerebrovascular accident (within 6 months before signing informed consent), myocardial infarction (within 6 months before signing informed consent), Unstable angina, congestive heart failure with NYHA class III or IV, or severe arrhythmias that cannot be controlled with medication or have a potential impact on study treatment; ECG results showing clinically significant abnormalities or QTcF ≥480 ms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with DLT at a Given Dose Level | 28 days
  Number of Subjects with DLT at a Given Dose Level（Low/Medium/High). A dose limiting toxicity (DLT) is defined as the hAESCs-related adverse event (AE) greater level than 3（including grade 3) that occurs during the DLT period, graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Maximum Tolerated Dose (MTD) | 28 days
  The Maximum Tolerated Dose (MTD) of hAESCs. The MTD is defined as the previous lower dose in the dose group in which ≥ 2/6 subjects developed DLT during the DLT observation period after infusion of hAESCs injection.
Incidence of adverse events | 100 days
  Incidence of adverse events (AEs), serious adverse events (SAEs), adverse events of special interest (AESIs).

SECONDARY OUTCOMES:
Overall response rate (ORR) | 100 days
  Overall response rate (ORR) after hAESCs injection infusion. ORR rate: the proportion of the total number of subjects who obtained CR, VGPR or PR after receiving study treatment to the total number of evaluable subjects.
Complete response (CR) rate | 100 days
  Complete response rate after hAESCs injection infusion. CR rate: the proportion of the total number of subjects who received a CR after receiving treatment to the total number of evaluable subjects.
Very good partial response (VGPR) rate | 100 days
  Very good partial response (VGPR) rate after hAESCs injection. VGPR rate: the proportion of the total number of subjects who received VGPR after receiving treatment to the total number of evaluable subjects.
Treatment ineffective rate | 100 days
  Treatment ineffective rate after hAESCs injection. Treatment ineffective rate: the proportion of the total number of participants who received NR or PD after receiving treatment to the total number of evaluable subjects.
Overall survival (OS) | 2 years
  Overall survival (OS) after infusion of hAESCs injection. OS: It refers to the time which begins at the start of treatment and up to the time of death.

OTHER OUTCOMES:
Maximum Plasma Concentration (Cmax) | 100 days
  The maximum plasma concentration will be obtained by PK analysis
Time to peak drug concentration (Tmax) | 100 days
  The time to peak drug concentration (Tmax) will obtained by PK analysis
T1/2(Half-Life) | 100 days
  The T1/2 will obtained by PK analysis
Area Under the Curve (AUC） | 100 days
  The Area Under the Curve (AUC) will obtained by PK analysis
The amount of IgM | 100 days
  The immunogenicity test of this product is aimed at the measurement of anti-drug antibodies after medication, including the measurement of IgM in vivo.
The amount of IgG | 100 days
  The immunogenicity test of this product is aimed at the measurement of anti-drug antibodies after medication, including the measurement of IgG in vivo.